CLINICAL TRIAL: NCT01873833
Title: Phase II Trial of Metronomic Capecitabine and Cyclophosphamide With Lapatinib and Trastuzumab in Patients With HER2 Positive Metastatic Breast Cancer Who Have Progressed on a Previous Trastuzumab-Based Regimen
Brief Title: Capecitabine, Cyclophosphamide, Lapatinib Ditosylate, and Trastuzumab in Treating Patients With HER2-Positive Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1B-12-10; NCI-2013-01086 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA014089 (NIH)
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: HER2-positive Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Cyclophosphamide; Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine; Trastuzumab; Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, lapatinib ditosylate, trastuzumab) (Experimental): Patients receive capecitabine by mouth (PO) every day (QD), cyclophosphamide PO QD, and lapatinib ditosylate PO QD on days 1-21 and trastuzumab IV on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: capecitabine; Drug: cyclophosphamide; Drug: lapatinib ditosylate; Biological: trastuzumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: capecitabine — Given PO
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Drug: cyclophosphamide — Given PO
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: lapatinib ditosylate — Given PO
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; Monoclonal antibody (MOAB) HER2; MOAB HER2
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well capecitabine, cyclophosphamide, lapatinib ditosylate, and trastuzumab work in treating patients with human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer. Drugs used in chemotherapy, such as capecitabine and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving capecitabine and cyclophosphamide daily may kill more tumor cells. Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for growth. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of the tumor to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving capecitabine, cyclophosphamide, lapatinib ditosylate, and trastuzumab together may be an effective treatment for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the progression free survival (PFS).

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate (ORR).

II. To evaluate the clinical benefit rate (CBR; complete response, partial response, and stable disease for >= 24 weeks).

III. To estimate the overall survival (OS).

IV. To assess the safety and tolerability.

OUTLINE:

Patients receive capecitabine orally (PO) once daily (QD), cyclophosphamide PO QD, and lapatinib ditosylate PO QD on days 1-21 and trastuzumab intravenously (IV) on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HER2-positive metastatic breast cancer
* HER2 overexpression of tumor by either immunohistochemistry (IHC) or fluorescence in situ hybridization (FISH); tumors tested by IHC must be 3+ positive; tumors tested by FISH must have a ratio of HER2: chromosome enumeration probe (CEP)17 > 2.0; when both tests are performed, the FISH result must be positive
* Prior trastuzumab use in the adjuvant or metastatic setting
* No more than two prior cytotoxic chemotherapeutic regimens for metastatic breast cancer. In addition, prior Trastuzumab emtansine (TDM-1, Kadcyla) is allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 9 g/dL
* Bilirubin =< 1.5 x upper limit of normal (ULN)
* Serum creatinine =< 1.5 x ULN or calculated creatinine clearance >= 60 ml/min
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN
* Fully recovered from toxicity due to prior therapy
* Capable of understanding the informed consent and complying with the protocol and signed the informed consent document prior to any study-specific screening procedures or evaluations being performed
* Must be able to swallow pills
* May have either measurable or non-measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Sexually active participants must agree to use a medically accepted barrier method of contraception (i.e. male condom or female condom) during the course of the study and for 3 months following discontinuation of study treatments; for participants of childbearing potential, a barrier method and a second method of contraception must be used
* Participants of childbearing potential must have a negative pregnancy test at screening and enrollment; participants of childbearing potential are defined as premenopausal females capable of becoming pregnant, i.e. females who have had any evidence of menses in the past 12 months with the exception of those who had prior hysterectomy (oophorectomy or surgical sterilization); however, women who have been amenorrheic for >= 12 months are still considered to be of childbearing potential if the amenorrhea is possibly due to any other cause including prior chemotherapy, antiestrogens, or ovarian suppression

Exclusion Criteria:

* Prior treatment with capecitabine or lapatinib
* Radiation therapy within 2 weeks before the first dose of study treatment
* Hormonal therapy within 2 weeks before the first dose of study treatment
* Cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) within 3 weeks before the first dose of study treatment
* Biologic therapy (including antibodies [other than trastuzumab], immune modulators, cytokines) within 4 weeks before the first dose of study treatment; Note: there is no washout period required for trastuzumab
* Any other type of investigational agent within 4 weeks before the first dose of study treatment
* Major surgery, or not recovered from major surgery within 4 weeks before the first dose of study treatment
* Untreated, symptomatic, or progressive brain metastases; participants must have no radiographic or other signs of progression in the brain for >= 1 month after completion of local therapy; any corticosteroid use for brain metastases must have been discontinued without the subsequent appearance of symptoms for >= 4 weeks prior to first study treatment
* Uncontrolled significant intercurrent illness that would preclude the patient from study participation per investigator assessment
* Left ventricular ejection fraction (LVEF) =< 50% as documented by multi gated acquisition scan (MUGA) or echocardiogram performed within 28 days prior to the first study treatment
* Currently receiving anticoagulation with therapeutic doses of warfarin (low-molecular weight heparin is permitted)
* Pregnant or breastfeeding
* Known to be positive for the human immunodeficiency virus (HIV) (a test for HIV at screening is not required)
* Have acute or currently active/requiring anti-viral therapy hepatic or biliary disease (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Previously identified allergy or hypersensitivity or intolerance to components of the study treatment formulation (cyclophosphamide, capecitabine, lapatinib [lapatinib ditosylate], trastuzumab)
* Any other diagnosis of malignancy or evidence of malignancy (except non-melanoma skin cancer, in-situ carcinoma of the cervix) within 2 years prior to screening for this study
* Unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07-29 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darcy V Spicer, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began recruiting in July 2013 and ended May 2017. Subjects were recruited from Los Angeles County + University of Southern California (LAC+USC) Healthcare Network and the Keck Medical Center of USC, Norris Comprehensive Cancer Center in Los Angeles, California.
Pre-assignment Details: There were no pre-assignment criteria. All subjects were given the same treatment.
Groups:
- Treatment (Chemotherapy, Lapatinib Ditosylate, Trastuzumab): Patients receive capecitabine PO QD, cyclophosphamide PO QD, and lapatinib ditosylate PO QD on days 1-21 and trastuzumab IV on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  capecitabine: Given PO
  cyclophosphamide: Given PO
  lapatinib ditosylate: Given PO
  trastuzumab: Given IV
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Lapatinib Ditosylate, Trastuzumab)
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Chemotherapy, Lapatinib Ditosylate, Trastuzumab): Patients receive capecitabine by mouth (PO) everyday (QD), cyclophosphamide PO QD, and lapatinib ditosylate PO QD on days 1-21 and trastuzumab IV on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  capecitabine: Given PO
  cyclophosphamide: Given PO
  lapatinib ditosylate: Given PO
  trastuzumab: Given IV
  laboratory biomarker analysis: Correlative studies
Arm/Group | Treatment (Chemotherapy, Lapatinib Ditosylate, Trastuzumab)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Scale: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; 5 = Dead
  Participants
    Status 0 | 4
    Status1 | 6
Breast cancer stage at diagnosis [Count of Participants; unit: Participants] — Staging was based on the American Joint Committee on Cancer (AJCC) 7th edition, with stage I having the best prognosis and stage IV having the worst prognosis.
  Participants
    II | 5
    III | 3
    IV | 2
Cancer Histologic Type (from surgical excision) [Count of Participants; unit: Participants]
  Ductal Infiltrating Carcinoma | 10
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as duration of time from the first dose of study drug to the first documentation of Progressive Disease (PD) by investigator assessment using RECIST 1.1 or death on study due to any cause on or before the data cutoff date, whichever occurred first. PD: >=20% increase (>=5 mm absolute increase) in the sum of target lesion measurements, compared to the smallest sum on study (including baseline), or unequivocal progression of non-target lesions, evaluated as a whole, such that it is clear that treatment has failed and disease is progressing, regardless of the status of the target lesions.
Time Frame: From study entry to the date of first documented disease progression (assessed every 6 weeks) or death due to any cause, whichever came first, approximately 63 months.
Population: All participants were included in the analysis. Statistical analysis was not performed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Chemotherapy, Lapatinib Ditosylate, Trastuzumab)
Number analyzed (Participants) | 10
months | 13.7 [2.6 to 16.6]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) is complete response (CR) + partial response (PR) recorded from study entry until disease progression based on RECIST v1.1 criteria. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: From study entry until disease progression/recurrence (maximum duration: 351 weeks)
Population: All patients were included in the analysis. Statistical analysis was not performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Lapatinib Ditosylate, Trastuzumab)
Number analyzed (Participants) | 10
Participants | 4

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Participants with a best response of CR, PR, or stable disease (SD) sustained for ≥24 weeks, as assessed using RECIST v1.1. CR: Disappearance of all non-nodal target and non-target lesions, including target and non-target lymph nodes reduction to <10 mm in short axis. PR: >=30% decrease in sum of diameters of target lesions, compared to the sum at baseline. SD: Neither PR nor progression of disease (PD) criteria met. SD follow PR only when sum increases by less than 20% from the nadir, but previously seen 30% decrease from baseline no longer hold. PD: >=20% increase (>=5 mm absolute increase) in the sum of target lesion measurements, compared to the smallest sum on study (including baseline), or unequivocal progression of non-target lesions, evaluated as a whole, such that it is clear that treatment has failed and disease is progressing, regardless of the status of the target lesions.
Time Frame: From study entry until the date of the first documented disease progression of date of death whichever came first, assessed for approximately 351 weeks
Population: All patients were included in the analysis. Statistical analysis was not performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Lapatinib Ditosylate, Trastuzumab)
Number analyzed (Participants) | 10
Participants | 7

4. Secondary Outcome: Overall Survival (OS)
Description: OS is the duration from study entry to death. Participants last known to be alive are censored at date of last contact.
Time Frame: From study entry until death from any cause or date of last contact (up to 70 months)
Population: All enrolled patients were included. Statistical analysis was not performed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Chemotherapy, Lapatinib Ditosylate, Trastuzumab)
Number analyzed (Participants) | 10
Months | 29.6 [11.8 to 81.9]

5. Secondary Outcome: Number of Participants With Any Adverse Events as a Measure of Safety and Tolerability
Description: Assessment based on CTCAE version 4.0 toxicity criteria. For the detailed list of adverse events see the adverse event module.
Time Frame: ****Time Frame: Adverse events were collected from first dose of study treatment up to 30 days after last dose of treatment, up to 63 months (number or treatment given ranged from 2 cycles to 85 cycles).
Population: All patients enrolled are included
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Lapatinib Ditosylate, Trastuzumab)
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning cycle 1 and continued throughout the study until 30 days after the last dose, up to 63 months.
Description: Adverse events (AE) graded according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0
Arm/Group | Treatment (Chemotherapy, Lapatinib Ditosylate, Trastuzumab)
All-Cause Mortality (participants affected / at risk) | 5/10
Serious Adverse Events (participants affected / at risk) | 5/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Chemotherapy, Lapatinib Ditosylate, Trastuzumab) (N=10)
10047700 - Vomiting (Gastrointestinal disorders) | 3
10016256 - Fatigue (General disorders) | 2
10034016 - Paronychia (Infections and infestations) | 1
10047900 - Weight loss (Investigations) | 3
10020639 - Hyperglycemia (Metabolism and nutrition disorders) | 1
10028411 - Myalgia (Musculoskeletal and connective tissue disorders) | 1
10054524 - Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
10002218 - Anaphylaxis (Immune system disorders) | 1
Death NOS (General disorders) | 5 — Death due to progressive disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Chemotherapy, Lapatinib Ditosylate, Trastuzumab) (N=10)
10002272 - Anemia (Blood and lymphatic system disorders) | 5
10008481 - Chest pain - cardiac (Cardiac disorders) | 1
10047340 - Vertigo (Ear and labyrinth disorders) | 1
10047848 - Watering eyes (Eye disorders) | 4
10000081 - Abdominal pain (Gastrointestinal disorders) | 9
10050068 - Edema limbs (General disorders) | 10
10019805 - Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 — Pain or discomfort in the area of the liver
Paronychia (Infections and infestations) | 3
10006504 - Bruising (Injury, poisoning and procedural complications) | 3
10001551 - Alanine aminotransferase increased (Investigations) | 7
10002646 - Anorexia (Metabolism and nutrition disorders) | 6
10003239 - Arthralgia (Musculoskeletal and connective tissue disorders) | 7
10013911 - Dysgeusia (Nervous system disorders) | 5
10002855 - Anxiety (Psychiatric disorders) | 5
10038359 - Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — Burning feeling when urinating, no infection.
10046937 - Vaginal pain (Reproductive system and breast disorders) | 1
10011224 - Cough (Respiratory, thoracic and mediastinal disorders) | 7
10037087 - Pruritus (Skin and subcutaneous tissue disorders) | 10
10020772 - Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT01873833/Prot_SAP_000.pdf